CLINICAL TRIAL: NCT05279677
Title: Phase II, Single-arm Study of FMT Combined With Immune Checkpoint Inhibitor and TKI in the Treatment of Colorectal Cancer Patients With Advanced Stage
Brief Title: FMT Combined With Immune Checkpoint Inhibitor and TKI in the Treatment of CRC Patients With Advanced Stage
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Vice director of Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3157
Record Dates: First submitted 2022-03-05; First posted 2022-03-15 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Neoplasms Malignant
Keywords: Gastrointestinal Microbiome
MeSH Terms: conditions — Colonic Neoplasms | interventions — Fecal Microbiota Transplantation; sintilimab; HMPL-013

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FMT (Experimental): Fecal microbiota transplantation plus Sintilimab and Fruquintinib
  Interventions: Drug: Fecal microbiota transplantation plus Sintilimab and Fruquintinib

INTERVENTIONS:
Drug: Fecal microbiota transplantation plus Sintilimab and Fruquintinib — Microbiota capsules containing 1g gut microbiota, po d1-3 before anti-tumor treatment, total for 8 cycles.
  Sintilimab 200mg iv, q3w. Fruquintinib 5mg po d1-14, q3w.

SUMMARY:
A single-arm, phase II study was designed to evaluate the efficacy and safety of fecal microbiota transplantation plus Sintilimab and Fruquintinib as the later line treatment in colorectal patients with advanced stages.

DETAILED DESCRIPTION:
The combination of regorafenib plus nivolumab had already presented a manageable safety profile and encouraging antitumor activity in patients with mCRC as the REGONIVO trail reported. While additional investigations showed limited ORRs between 7%-33% as third or later line treatement in mCRC. Gut microbiota modulation, with the aim to reverse established microbial dysbiosis, is a novel strategy for the treatment of CRC. The individualized gut microbiome transplantation may further imrpove the efficacy of the combination therapy of CPI and TKI. Thus, a single-arm, phase II study was designed to evaluate the efficacy and safety of FMT plus Sintilimab and Fruquintinib as the later line treatment in CRC patients with advanced stages.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form.
* Metastatic or locally advanced colorectal adenocarcinoma unresectable or unfit for radical radiochemotherapy confirmed by pathology or cytology.
* Microsatellite stable or pMMR patients failed standard treatment, including platinum, irinotecan, fluorouracil and Bevacizumab (Ras and BRAF wt patients should recived Cetuximab).
* Patients have at least one lesion could be evaluated by RECIST v1.1 or mRECIST.
* The Eastern Cooperative Oncology Group (ECOG) performance status score was 0 or 1.
* The life expectancy is more than 3 months.
* Good organ function:

Blood routine: hemoglobin ≥90g/L, white blood cell ≥3.0×10^9/L, neutrophil ≥1.5×10^9/L, platelet ≥100×10^9/L; Renal function: creatinine≤1.5×upper limit of normal (UNL) or creatinine clearance ≥60ml/min; Liver function: total bilirubin (TBIL)≤1.5×upper limit of normal (UNL); ALT≤2.5×UNL, AST≤2.5×UNL, ALT≤5×UNL and AST≤5×UNL for patients with liver metastasis.

Exclusion Criteria:

* Have received any anti-PD-1, anti-PD-L1/L2 antibodies, anti-CTLA-4 antibodies and other immunotherapy in the past.
* Have received any TKI therapy in the past.
* Clinically significant ascites.
* Known to have allergic reactions to any ingredients or excipients of experimental drugs.
* Have received any antibiotics within 28 days before the first medication or any probiotics or prebiotics within 14 days before the first medication.
* Radiotherapy, RFA, interventional therapy or surgery were performed within 28 days before the first medication (except for previous diagnostic biopsy).
* Other active malignant tumors, excluding those who have been disease free for more than 5 years or in situ cancer considered to have been cured by adequate treatment.
* Brain metastasis or meningeal metastasis has been confirmed. Patients with neurological symptoms should receive brain CT / MRI examination to exclude metastasis.
* Patients who is suffering from intestinal obstruction, gastrointestinal bleeding, pulmonary fibrosis or interstitial pneumonia, renal failure, liver failure or cerebrovascular disease.
* Diabetes was not controlled, defined as HbA1c > 7.5% after anti-diabetic drugs or hypertension was not controlled, defined as systolic / diastolic blood pressure > 140 / 90 mmHg after antihypertensive drug.
* Myocardial infarction, severe/unstable angina, New York Heart Association (NYHA) class III or IV congestive heart failure in the past 12 months.
* Known to be infected with human immunodeficiency virus (HIV), have acquired immunodeficiency syndrome (AIDS) related diseases, have active hepatitis B or hepatitis C.
* Suffering from autoimmune diseases or history of organ transplantation requiring immunosuppressive therapy.
* May increase the risk associated with participation in the study or administration of the study drug or mental illness that may interfere with the interpretation of research results.
* Pregnant women (determined by serum human chorionic gonadotropin [hCG]) or lactating women, or plan to conceive during the treatment period, 2 months after cetuximab treatment and 6 months after capecitabine treatment. Women of childbearing age with positive or no pregnancy test at baseline. Women of childbearing age or sexually active men were not willing to use contraception during the study period, at least 2 months after cetuximab treatment and 6 months after capecitabine treatment. Postmenopausal women must be amenorrhea for at least 12 months to be considered infertile.
* There are other serious diseases that the researchers believe patients cannot be included in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 2 years
  Objective Response Rate

SECONDARY OUTCOMES:
OS | Up to 2 years
  Overall Survival
PFS | Up to 2 years
  Progression Free Survival
Adverse events | Up to 2 years
  Safety and tolerance

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No